CLINICAL TRIAL: NCT01962428
Title: Randomized Trial of Different Loading Dose of Ticagrelor for Antiplatelet Effect in Patients With Non -ST-segment Elevation ACS Undergoing Percutaneous Coronary Intervention
Brief Title: Different LD of Ticagrelor for Antiplatelet Effect in Patients With Non-ST-segment Elevation ACS Undergoing PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0214
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2015-12

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome
Keywords: ticagrelor; loading dose; non-ST-segment elevation acute coronary syndromes; percutaneous coronary intervention; the antiplatelet effects; bleeding events; major adverse cardiac events
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high loading dose of ticagrelor (Experimental): Patients will receive ticagrelor 360mg loading dose, then 90mg bid maintenance dose starting 12 hours after loading dose.
  Interventions: Drug: ticagrelor
- conventional loading dose of ticagrelor (Active Comparator): Patients will receive ticagrelor 180mg loading dose, then 90mg bid maintenance dose starting 12 hours after loading dose.
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: ticagrelor — Patients will receive ticagrelor 360mg loading dose or 180mg loading dose , then 90mg bid maintenance dose starting 12 hours after loading dose.
  Other Names: Brilinta

SUMMARY:
It is designed to test the hypothesis that high loading dose(360mg) ticagrelor versus conventional loading dose(180mg) will result in a higher inhibition of platelet aggregation(IPA) without increasing the bleeding events.

DETAILED DESCRIPTION:
After providing written informed consent, all patients will be randomized to receive ticagrelor 360mg or 180mg loading dose(LD),then 90mg bid maintenance dose starting 12 hours after LD.PCI will performed in 2h-72h after they are given the loading dose.All patients should receive acetylsalicylic acid (ASA) 75 to 100 mg daily unless intolerant.IPA at 0, 0.5, 1, 2, 8, 24h after the loading dose of ticagrelor will be measured. CK-MB, troponin I, myoglobin, CRP will be detected at 0h, before PCI, 8h after PCI, 24h after PCI. ECG will be conducted at 0h and within 24h after PCI. Patients returned 28 days for follow-up visits after the loading dose of ticagrelor, documented any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Male or non-pregnant female; aged from 18 to 80 years old.
* Patients with non-ST-segment elevation acute coronary syndromes who were scheduled to undergoing PCI.

Exclusion Criteria:

* Any contraindication against the use of ticagrelor.
* On treatment with a P2Y12 receptor antagonist in past 30 days.
* Known allergies to aspirin or ticagrelor.
* On treatment with oral anticoagulant (Vitamin K antagonists, dabigatran, rivaroxaban).
* Known blood dyscrasia or bleeding diathesis.
* ST-segment elevation acute myocardial infarction.
* Non-ST segment elevation acute coronary syndrome with high-risk features warranting emergency coronary angiography.
* Left ventricular ejection fraction ≤30%; renal failure with creatinine 3 mg/dl; history of liver disease; an increased risk of bradycardia, and concomitant therapy with drugs interfering with CYP3A4 metabolism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huiliang Liu, Doctor, Principal Investigator — Department of Cardiology of General Hospital of Chinese People's Armed Police Forces
Locations (2):
- China (2):
  - General Hospital of Chinese People's Armed Police Forces, Beijing, Beijing Municipality
  - General Hospital of Chinese People's Armed Police Forces, Beijing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 278 patients were recruited at 8 centers in Beijing and allocated into two groups using block randomization: a high LD group (360 mg) and a conventional LD group (180 mg).
Pre-assignment Details: Patients excluded(n=564)
Period: Overall Study
Arm/Group | High Loading Dose of Ticagrelor | Conventional Loading Dose of Ticagrelor
Started | 139 | 139
Completed | 129 | 133
Not Completed | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Loading Dose of Ticagrelor | Conventional Loading Dose of Ticagrelor | Total
Number analyzed (Participants) | 129 | 133 | 262
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 80 | 155
  >=65 years | 54 | 53 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (9.47) | 58.8 (10.26) | 59.2 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 45 | 85
  Male | 89 | 88 | 177
Region of Enrollment [Number; unit: participants]
  China | 129 | 133 | 262

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Index(PRI) Measured by VASP-P
Description: Vasodilator-stimulated phosphoprotein(VASP) phosphorylation, a measure of P2Y12 receptor reactivity, was determined by flow cytometry with the use of the Platelet VASP-FCM Kit (Stago, France)and recorded as the platelet reactivity index (PRI).
Time Frame: 2 hours after the loading dose of ticagrelor
Measure: Median (Inter-Quartile Range); unit: percentage of 100
Arm/Group | Conventional Loading Dose of Ticagrelor | High Loading Dose of Ticagrelor
Number analyzed (Participants) | 133 | 129
percentage of 100 | 16.7 [4.3 to 21.3] | 12.2 [9.3 to 32.3]

2. Secondary Outcome: Platelet Reactivity Index (PRI) Measured by VASP-P
Time Frame: 0.5hour,1hour,8hours,24hours after the loading dose of ticagrelor
Reporting Status: Not Posted

3. Secondary Outcome: Bleeding Events
Time Frame: follow-up for 28 days after the loading dose of ticagrelor
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Conventional Loading Dose of Ticagrelor | High Loading Dose of Ticagrelor
Serious Adverse Events (participants affected / at risk) | 3/139 | 5/139
Other Adverse Events (participants affected / at risk) | 15/139 | 19/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Conventional Loading Dose of Ticagrelor (N=139) | High Loading Dose of Ticagrelor (N=139)
aortic dissection (Cardiac disorders) | 1 (1) | 0/129 (0) — Complication of aortic dissection emerged when the patient underwent PCI .
pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) — patient was diagnosed pericardial effusion, pericardialtamponade after LAD-PCI, his vital signs were unstable.Antiplatelet drugs such as ticagrelor , aspirin were withdrawn.
death (Cardiac disorders) | 1 (1) | 1 (1)
AMI (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastrorrhagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
failure of PCI (Cardiac disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Loading Dose of Ticagrelor (N=139) | High Loading Dose of Ticagrelor (N=139)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days